CLINICAL TRIAL: NCT04700475
Title: Effect of Low Level Laser Therapy on Prevention of Radiotherapy Induced Xerostomia in Cancer Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nada Yousef (Other)
Responsible Party: Sponsor-Investigator, Nada Yousef, Assistant lecturer of physical therapy, cairouniversity, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P.T.REC/012/002269
Record Dates: First submitted 2020-09-29; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Head and Neck Cancer
Keywords: Low level laser; Xerostomia; Radiotherapy; Head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia | interventions — Low-Level Light Therapy; citric acid, deuterium oxide solution

STUDY DESIGN:
Intervention Model Description: In the study, 2 groups of patients will participate First, study group will recieve low level laser on major salivary glands and usual medications.
  Second, control group will recieve usual medications. Second, control
Who Masked: Participant, Care Provider, Investigator
Masking Description: The participants are head and neck cancer patients recieving radiotherapy. The care provider are oncologist and nursing stuff. The investigator is phsical therapist (my self)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): Laser group composes of thirty patients who will receive low level laser three times a week, on alternate day (48h interval) Laser therapy will be initiated before the first radiotherapy session and ended after the last session, totaling 21 sessions
  Interventions: Device: low level laser; Drug: citric acid solution
- Control group (Other): control group composes of thirty patients will be treated with 15mL of a 2% citric acid solution applied as a mouth rinse for 30 sec
  Interventions: Drug: citric acid solution

INTERVENTIONS:
Device: low level laser — Laser will be performed with a GaAlAs diode laser at a wavelength of 808 nm, 100-mW output power, laser beam area of 0.03 cm2, and in continuous wave mode, three times a week, on alternate days. Laser therapy will be initiated before the first radiotherapy session and ended after the last session, totaling 21 sessions.
  The total energy per session (56 J) will be divided into 14 irradiation points, as marked on the overlying skin (Fig.2). Each irradiation point received a dose of 4 J over an irradiation time of 40 s.
  With exclusion of tumor area or area of removed tumor laser will be applied as following:
  • Extra oral application: The laser will be used extraorally at eight points in the parotid glands (bilaterally, four points in each gland), at four points in the submandibular glands (bilaterally, two points in each gland
  • Intraoral application: The will be used intraorally at two points in the sublingual glands bilaterally, one point in each gland .
  Other Names: cold or non invasive laser
  Arms: Laser group
Drug: citric acid solution — citric acid solution applied as a mouth rinse

SUMMARY:
The purpose of the study is to evaluate the effectiveness of low level laser on radiotherapy induced xerostomia to improve oral function and decrease oral complication due to hyposalivation and thus enhancing survival.

DETAILED DESCRIPTION:
In this part of the study, the materials and methods will be presented under the following headings: subjects, equipment, procedures of the study and the statistical procedures.

1. Subjects:

   Sixty patients who have head and neck cancer (oral cavity, pharynx, larynx, or occult primary tumor) submitted to conventional 3D radiotherapy, with irradiation fields necessarily encompassing all major salivary glands. The total dose ranged from 66 to 70 Gy, given in fractions of 2 Gy/day selected randomly from Nuclear medicine department, Oncology institute, Mansoura University.

   These patients will be divided randomly into two groups of equal number, thirty patients for each group.

   Group A: (Laser group) This group of patients composes of thirty patients who will receive GaAlAs laser three times a week, on alternate day (48h interval) Laser therapy will be initiated before the first radiotherapy session and ended after the last session, totaling 21 sessions (Fernanda A. S.G. et al., 2016).

   Group B :( Control group) This group of patients composes of thirty patients will be treated with 15mL of a 2% citric acid solution applied as a mouth rinse for 30 sec (Bozana Loncar, D.M.D. et al., 2010) .

   The criteria of Patients selection :
2. Equipment used:

1-Therapeutic equipment: Laser therapy will be performed with an GaAlAs laser

2- Evaluation tools:

* Unstimulated and stimulated saivery flow rate.
* Salivery immunoglobin A (sIgA) concentration in unstimulated saliva
* The 11-item modified Xerostomia Inventory-Dutch questionnaire version 22.

ELIGIBILITY:
Inclusion Criteria:

* - Age range between 25-55 years.
* All patients included in the study established HNC and will receive radiotherapy encompassing major salivary glands accompanied or not by surgery.
* All patients enrolled to the study will have their informed consent.
* Both genders will participate in the study.
* All the patients were examined medically by oncologist

Exclusion Criteria:

* - Diabetes mellitus,
* Autoimmune diseases as sjorgen syndrome by established diagnosis criteria.
* Infectious diseases
* Collagen diseases, as were those with incipient tumors (stage T1 or T2) limited to the larynx, as well as those with trismus (reduced mouth opening capacity) due to surgical sequelae.
* xerostomic drugs (antiretroviral medications, antihistamines, anticholinergics, antihypertensives, decongestants, narcotic analgesics, tricyclic antidepressants)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-04 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Unstimulated and stimulated salivary flow rate. | 7 weeks
  For the assessment of salivary flow rate, unstimulated and stimulated sialometry tests will be performed before the first radiotherapy session and after completion of laser programe.
  As salivary secretion fluctuates between minimal and maximal rates during the day, it is important to assess the salivary secretion consistently at an established time of the day, in order to properly examine the evolution of the condition and its treatment in every patient.
  The normal flow rate for unstimulated, "resting" whole saliva is 0.3 to 0.5 ml/min.; for stimulated saliva, 1 to 2 ml/min. Values less than 0.1 ml/min. are typically considered xerostomic, although reduced flow may not always be associated with complaints of dryness

SECONDARY OUTCOMES:
Salivary immunoglobin A (sIgA) concentration in unstimulated saliva. | 7weeks
  The samples of unstimulated whole saliva will be frozen and stored at -20°C until used for sIgA determination. sIgA concentrations were measured by using commercially available indirect competitive enzyme immunoassay kit (Salivary SIgA EIA kit, Salimetrics).
  The quantities of salivary IgA secreted in 5 minutes will be calculated by taking in account sIgA concentrations and volumes of unstimulated saliva secreted in 5 minutes.

OTHER OUTCOMES:
The 11-item modified Xerostomia Inventory-Dutch questionnaire version | 7weeks
  The XI is an 11-item summated rating scale that was developed to measure the severity of dry mouth symptoms. The final score ranges from 5 to 55, with higher scores indicating more severe symptoms. A decrease in XI scores of 6 points or more between pre- and post-treatment assessments will be considered clinically significant.
  The mean dry mouth score and the correlation between dry mouth score and salivary flow rate will be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No